CLINICAL TRIAL: NCT06681805
Title: Role of Prophylactic Mirtazapine and Different Doses of Intrathecal Morphine in Preventing Nausea and Vomiting After Cesarean Section: A Randomized Controlled Trial
Brief Title: Prophylactic Mirtazapine and Different Doses of Intrathecal Morphine in Preventing Nausea and Vomiting After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Basma Mohamed Ghoniem, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelshiekh University, Kafrelshiekh, Egypt, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR752/7/24
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Prophylactic; Mirtazapine; Intrathecal; Morphine; Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Mirtazapine; Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Groups I (Experimental): Patients received 30mg of oral mirtazapine one hour before surgery plus 10 mg of bupivacaine 0.5% along with 0.2 mg of morphine.
  Interventions: Drug: Mirtazapine + Bupivacaine + Morphine
- Groups II (Experimental): Patients received 30mg of oral mirtazapine one hour before surgery plus 10 mg of bupivacaine 0.5%, along with 0.1 mg of morphine.
  Interventions: Drug: Mirtazapine + Bupivacaine + Morphine
- Groups III (Placebo Comparator): Patients received a placebo one hour before surgery plus 10 mg of bupivacaine 0.5%, along with 0.2 mg of morphine.
  Interventions: Drug: Placebo + Bupivacaine + Morphine
- Groups IV (Placebo Comparator): Patients received a placebo one hour before surgery plus 10 mg of bupivacaine 0.5%, along with 0.1 mg of morphine.
  Interventions: Drug: Placebo+ Bupivacaine + Morphine

INTERVENTIONS:
Drug: Mirtazapine + Bupivacaine + Morphine — Patients received 30mg of oral mirtazapine one hour before surgery plus 10 mg of bupivacaine 0.5% along with 0.2 mg of morphine.
  Arms: Groups I
Drug: Mirtazapine + Bupivacaine + Morphine — Patients received 30mg of oral mirtazapine one hour before surgery plus 10 mg of bupivacaine 0.5%, along with 0.1 mg of morphine.
  Arms: Groups II
Drug: Placebo + Bupivacaine + Morphine — Patients received a placebo one hour before surgery plus 10 mg of bupivacaine 0.5%, along with 0.2 mg of morphine.
  Arms: Groups III
Drug: Placebo+ Bupivacaine + Morphine — Patients received a placebo one hour before surgery plus 10 mg of bupivacaine 0.5%, along with 0.1 mg of morphine.
  Arms: Groups IV

SUMMARY:
The aim of this work was to evaluate the role of prophylactic mirtazapine and different doses of intrathecal morphine in preventing nausea and vomiting.

DETAILED DESCRIPTION:
It is common practice to provide intrathecal morphine to alleviate postoperative pain because of its powerful and long-lasting analgesic effects. Mirtazapine is a noradrenergic and specific serotonergic antidepressant. It is anxiolytic by its antagonist of the 5HT2 receptor and is strongly sleep-inducing. Its antagonist at 5-hydroxytryptamine subtype 3 (5-HT3) receptor may help to prevent nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Scheduled for caesarean section under spinal anesthesia

Exclusion Criteria:

* Known hypersensitivity to mirtazapine.
* Gastrointestinal illness.
* Diabetes mellitus.
* Use of opioids or any medication with known antiemetic properties within 48 hours before surgery.
* Mental disorders.
* Spinal anesthesia contraindications.
* Taking antidepressants or antipsychotic medications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women scheduled for a cesarean section
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 24 hours postoperatively
  Incidence of postoperative nausea and vomiting was recorded at 3, 6, 12, 18, 24 hours postoperatively.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient was instructed about postoperative pain assessment with the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS was assessed at 0, 3, 6, 12, 18, 24 hours postoperatively.
Time to first rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to the first dose of pethidine administrated).
Total pethidine consumption | 24 hours postoperatively
  Rescue analgesia of pethidine 0.5μg/kg was given as a bolus if the numeric rating scale (NRS) > 3.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as itching, bradycardia, hypotension, pruritis, urinary retention, headache, respiratory depression, miosis, and seizures were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.